CLINICAL TRIAL: NCT01912092
Title: A NON-CONTROLLED PROSPECTIVE COHORT STUDY OF THE USE OF ASKINA® CALGITROL® PASTE + STANDARD OF CARE ON MILDLY INFECTED, NON-ISCHAEMIC DIABETIC FOOT ULCERS
Brief Title: Askina Calgitrol Paste Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPM-O-H-1205
Record Dates: First submitted 2013-07-25; First posted 2013-07-30 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Diabetic Foot Ulcer (DFU)
MeSH Terms: conditions — Diabetic Foot

ARMS (1):
- Askina Calgitrol Paste (Experimental)
  Interventions: Device: Askina Calgitrol paste

INTERVENTIONS:
Device: Askina Calgitrol paste

SUMMARY:
The purpose of this study is to assess the efficacy of Askina® Calgitrol® Paste in reducing local infection in subjects treated for mildly infected Diabetic Foot Ulcers (DFU) with Askina® Calgitrol® Paste.

ELIGIBILITY:
Inclusion Criteria:

* Subject older than 18 years old
* Provision of written consent by the subject themselves
* Subjects with a Texas stage I-B wound below the malleolus: superficial and infected (Wagner-Armstrong classification system).
* Subjects with a mildly infected wound according to the Infectious Diseases Society of America (IDSA).
* Size of wound >2 cm2.
* Absence of ischaemia of the lower limb as assessed by :

  1. Transcutaneous oxygen pressure (TcPO2) > 30 mmHg.
  2. Toe pressure > 50 mmHg.
  3. Ankle pressure > 70 mmHg.
* Capable of following Study instructions.
* Compliant with treatment and in particular with off-loading regime.
* Stable management of their diabetes as defined by an HbA1C (%) of 12%

Exclusion Criteria:

* Subjects who are <18 years old.
* Subjects with a documented sensitivity to alginates or silver.
* Subjects taking a medication or using a device comprising silver.
* Subjects already taking antibiotics before enrolment
* Subjects undergoing dialysis.
* Subjects using therapy known to be immune-compromising such as systemic anti-neoplastic drugs and/or systemic cortico-steriods.
* Pregnancy
* Breast-feeding
* Currently participating in another clinical trial, or who have participated in another clinical trial in the last 6 weeks or who have previously taken part in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Clinical signs of local infection (Presence of erythema, pain, tenderness, warmth or induration) | At day 0, day 2 and weekly in a period of a maximum of 6 weeks
  During each of the day 2 and weekly control visits, the investigator will observe the wound visually and assess it for signs of Clinical infection, using the Guidelines for Diabetic Foot Ulcer infection of the Infectious Diseases Society of America. The investigator will score the degree of infection of the wound according to a table adapted from the 8 items wound score for diabetic foot infections.
  In general, treatment with Askina Calgitrol Paste will be discontinued when local infection has resolved or when it was worsened since the last control visit. However, treatment of Askina Calgitrol Paste will continued after 4 weeks of treatment only if there are signs of improvement.
  The treatment period of Askina Calgitrol Paste will last a maximum of 6 weeks.

SECONDARY OUTCOMES:
Adverse events or Adverse device related event | At day 2 and weekly in a period of a maximum of 6 weeks
Evaluation of wound bed (necrosis, slough, granulation, epithelialisation) | At day 0, day 2 and weekly in a period of a maximum of 6 weeks
  It will be assessed visually by the investigator.
Ease of use of Askina Calgitrol Paste | Daily or at every change of dressing, in a period of a maximum of 6 weeks
  Ease of application and removal of dressing will be assessed by the subject/subject's relatives and the investigator using a rating scale of 1 (very easy) to 5 (very difficult). Dressing change at home will be evaluated in a patient diary by the patient or the carer and dressing changes in the clinic by the investigator.
Wound surface area | At day 0, day 2 and weekly in a period of a maximum of 6 weeks
  It will be measured by Visitrak Wound Measurement System at each clinic visit by the healthcare professional.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Diabetic Foot and metabolic diseases clinic, Milan
  - IRCCS Casa di Cura MultiMedica, Milan